CLINICAL TRIAL: NCT03732274
Title: Phase 1b/2a, Open Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of Vactosertib in Combination With Durvalumab in Patients With Advanced Non Small Cell Lung Cancer Who Progressed Following Platinum-based Chemotherapy
Brief Title: Phase 1b/2a, Open-label Study of Vactosertib in Combination With Durvalumab in Advanced NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedPacto, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-VAC-203
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation of TEW-7197 (Experimental): TEW-7197 will be administered orally for 5 days per week (5D/W) and Durvalumab administration.
  Interventions: Drug: TEW-7197

INTERVENTIONS:
Drug: TEW-7197 — TEW-7197 will be administered orally for 5 days per week (5D/W) at the same time in the morning and evening (BID) approximately 12 hours apart. Durvalumab will be administered as a dose of 1500 mg every 4weeks.
  Other Names: vactosetib

SUMMARY:
This is an open -label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of Vactosertib in Combination with durvalumab in patients advanced NSCLC who progressed following platinum-based chemotherapy.

DETAILED DESCRIPTION:
This is Phase 1b/2a, open label, multi-center study to assess safety, tolerability, pharmacokinetics and anti-tumor activity of vactosertib in combination with durvalumab in patients advanced NSCLC. This study has been designed to allow for an investigation of the optimal dose of vactosertib in combination with durvalumab. There are two parts to this study: Phase 1b, vactosertib dose-escalation study to determine the recommended phase 2 dose (RP2D) and Phase 2a, non-randomized parallel dose expansion study to confirm RP2D.

In the current dose-escalation (Phase 1b) study to determine RP2D, vactosertib dosing will begin at 100 mg BID for 5 days per week in combination with durvalumab 1500 mg, Q4W. According to the following dose escalation rule, 200 mg BID oral dose as maximum administered dose (MAD) will be administered in combination with durvalumab.

This phase 2a study is a study designed to evaluate the anti-tumor effects of vactosertib in combination with durvalumab in a total of 45 patients with PD-L1 positive advanced NSCLC who progressed following platinum-based chemotherapy (no prior immunotherapy)

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Age ≥19 years at the time of screening
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 at enrollment
4. Histological or cytological confirmation of advanced NSCLC who progressed following platinum-based chemotherapy.
5. If there is measurable disease based on RECIST 1.1 identified by the investigator at screening and there is at least one non-irradiated lesion suitable for selection as a target lesion according to RECIST 1.1 on imaging test, tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to the first dose.
6. No prior exposure to immune-mediated therapy including, but not limited to, other anti CTLA-4, anti-PD-1, anti-PD-L1, and anti programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines for treatment purpose.
7. In dose escalation phase, 6 DLT evaluable patients whose tumor cell PD-L1 expression less than 25% will be enrolled in each cohort. In dose expansion phase, 45 patients with confirmed PD-L1-positive NSCLC by using the Ventana SP263 IHC assay will be enrolled

   * Evaluation in newly acquired tumor tissue (preferred) or archival tissue (≤3 years old).
   * If the patient's PD-L1 status has already been assessed using Ventana SP263 assay, this test result can be used to assess eligibility for enrollment.
   * Note: A positive PD-L1 sample is measured using a defined cut-off based on ≥1% of tumor cells with membrane staining of any intensity for PD-L1.
8. All patients must be able to provide an available tumor sample collected within ≤3 years after the last anticancer therapies prior to screening. At least 25 patients enrolled in the dose expansion phase must be able to provide newly acquired tumor biopsy taken within 6 months prior to the first dosing. Tumor lesions used for newly acquired biopsies should not be target lesions, unless there are no other lesions suitable for biopsy, and only a core needle (not excisional/incisional) biopsy is allowed when biopsies are performed on target lesions as there is no other lesions suitable for biopsy. In patients with only one target lesion, biopsy for baseline tumor evaluation should be performed prior to the imaging test with an interval of at least 2 weeks after biopsy. Samples with limited tumor content and fine needle aspirate specimens are not acceptable. Specimens from metastatic bone lesions are typically unacceptable unless there is a significant soft tissue component. The tumor specimen quantity should be as sufficient as possible to allow for exploratory biomarker analyses and is preferred in formalin-fixed paraffin embedded blocks. An additional subsequent tumour biopsy will be performed on C2D3-6 or C2D10-13 only in patients who provide newly acquired tumor biopsy taken within 6 months prior to the first dosing. The same tumor lesion should be biopsied at all timepoints, if feasible, to avoid introduction of heterogeneity related to the site of tumor or metastasis.
9. Adequate organ and marrow function as defined below:

   * Hemoglobin ≥9.0 g/dL
   * Absolute neutrophil count ≥1.0 × 109 /L
   * Platelet count ≥75 × 109/L
   * Serum bilirubin ≤1.5 × the upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed enrollment in consultation with their physician.
   * ALT and AST ≤2.5 × ULN; for patients with hepatic metastases, ALT and AST ≤5 × ULN
   * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance (CL) >40 mL/min as determined by Cockcroft-Gault (using actual body weight)
10. Must have a life expectancy of at least 12 weeks
11. Body weight >30 kg
12. Male and/or female

Exclusion Criteria:

1. History of allogeneic organ transplantation.
2. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the Study Physician
   * Patients with celiac disease controlled by diet alone
3. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association [NYHA] Class III/IV), uncontrolled hypertension (≥150/90 mmHg), unstable angina pectoris, myocardial infarction (≤ 6 months prior to screening), clinically significant cardiac valvulopathy requiring treatment, uncontrolled cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
4. History of another primary malignancy except for

   * Malignancy tumors with low risk of recurrence treated with curative intent and with no known active disease ≥5 years before the first dose of IP Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease
5. History of leptomeningeal carcinomatosis
6. History of active primary immunodeficiency
7. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (HBV surface antigen [HBsAg] test positive), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody (anti-HBc) and negative of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only with negative HCV RNA measured by polymerase chain reaction.
8. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory test results coinciding with the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity expected not to be exacerbated by study treatment may be included only after consultation with the Study Physician.
9. In the case of brain metastases or spinal cord compression, patients with suspected brain metastases at screening should undergo a brain MRI (preferred) or CT test using IV contrast medium prior to study entry. Brain metastases will not be recorded as RECIST Target Lesions at baseline. Note: Patients whose brain metastases have been treated may participate provided they show radiographic stability defined as 2 brain imaging results, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least 4 weeks apart and show no evidence of intracranial progression. In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤10 mg/day of prednisone or its equivalent for at least 14 days prior to the start of treatment.
10. QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥450 ms in male and ≥470 ms in female
11. Known allergy or hypersensitivity to any of the study drugs or the study drug excipients Prior/concomitant therapy
12. Administration of the last dose of anticancer therapy (chemotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, or monoclonal antibodies) ≤ 3 weeks prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the medication administration schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by Sponsor and the Investigator. Concurrent use of following therapies is acceptable.

    * Hormonal therapy with gonadotropin-releasing hormone (GnRH) agonists or antagonists for prostate cancer
    * Hormone-replacement therapy or oral contraceptives
    * The situation in which a regulatory agency allows a regulatory agency approved tyrosine kinase inhibitor (TKI) is the case in which TKI is administered prior to a period of at least 7 days beginning on day 1 of the first cycle of the trial.Baseline scans must be obtained after discontinuation of prior TKIs, and registration criteria pertaining to adverse events related to prior anticancer therapies must be met.
    * The situation in which herbal therapy is allowed is when the herbal medicine has been administered at least one week prior to Day 1 of Cycle 1.
13. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks of the first dose of study treatment.
14. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
15. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of study drugs. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
17. The prohibited medications when using vactosertib are following (Refer to Appendix E);

    * The concurrent use of strong CYP3A4 inhibitors, including but not limited to grapefruit juice, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, voriconazole are not allowed in the study (The use of tropical drugs such as 2% ketoconazole cream, may be allowed when discussed with the Sponsor).
    * The concurrent use of potent CYP3A4 inducers, including but not limited to phenytoin, rifampin, and St. John's wort, are not allowed in the study.
    * Substances with a sensitive or narrow therapeutic range of CYP including but not limited to: efavirenz, theophylline, darunavir, dasatinib, everylimus, lopinavir, midazolam, sirolimus, ticagrella, astemizole, cisapride, cyclosporine, dihydroergotamine, ergotamine, sirolimus, tacrolimus, terfenadine
    * Drug use exclusively or mainly removed by UGT1A1 is not allowed in the study. Prior/concurrent clinical study experience
18. Participation in another clinical study with an investigational product administered in the last 30 days
19. Previous IP assignment in the present study
20. Concurrent enrollment in another clinical study, excluding an observational (non interventional) clinical study or during the follow-up period of an interventional study Other exclusions
21. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab or vactosertib, whichever is longer.
22. Judgment by the Investigator that the patient should not participate in the study if unlikely to comply with study procedures, restrictions, and requirements.
23. For genetics research study, the followings are excluded;

    * Previous allogeneic bone marrow transplant
    * Non-leukocyte-depleted whole blood transfusion within 120 days of genetic sample collection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 4 weeks
  To define the MTD

SECONDARY OUTCOMES:
Number of participants with treatment -related adverse events | From screening through study completion (up to 28 days after the last dose of Investigational Drug)
  To evaluate safety profile of TEW-7197 with regards to frequency, type,grade and seriousness and causality of treatment-related clinical and laboratory adverse events
Objective Response Rate (%) | every 2 cycles (each cycle is 28 days) and end of treatment (EOT) time point ,EOT is defined as within 30 days from the last dose of study medication by the protocol
  ORR of TEW-7197 in combination with durvalumab by RECIST v1.1
Pharmacokinetics (PK) of TEW-7197 | At cycle 1 (each cycle is 28 days)
  Peak Plasma Concentration of TEW-7197
Pharmadynamics of TEW-7197 | At cycle 1 ,3 (each cycle is 28days)
  Circulating cytokines including TGF-β1, PAI-1

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Heo, Study Director — MedPacto, Inc.
Locations (4):
- South Korea (4):
  - ChungBuk national university hospital, Chungju
  - National Cancer Center, Goyang-si
  - Yeonsei University Hospital, Seoul
  - The Catholic univ of korea st.vincent's hospital, Suwon